CLINICAL TRIAL: NCT04220177
Title: Prospective, Open-label, Multicenter, Non-randomized Clinical Study to Determine the Safety and Efficacy of SETA LATECBA Stent Graft for Endovascular Repair Therapy (EVAR) in Subjects With Abdominal Aortic Aneurysm (AAA).
Brief Title: Safety and Efficacy of the SETA LATECBA Stent Graft for EVAR in Subjects With AAA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Latecba S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SETALATECBACAN002
Record Dates: First submitted 2020-01-05; First posted 2020-01-07 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Intervention Model Description: Prospective, Open-label, Multicenter, Non-randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment arm (Experimental): SETA LATECBA Stent Grafts, are tube shaped implantable devices, delivered by balloon catheter system which are intended to the treatment of infrarenal AAA by sealing the affected areas, avoiding the bleeding or perfusion inside the aneurysm and restoring the normal hemodynamics in the affected vessels. The product family is composed by a set of endovascular stent grafts, that can be used alone or in combination, according to the treatment strategy, extension and complexity of the AAA. One aortic bifurcated stent graft, ABK SETA LATECBA model, is the aortic trunk and two straight iliac stent grafts, RIK SETA LATECBA model, are the connections to both iliac arteries.
  Interventions: Device: SETA LATECBA Stent Grafts

INTERVENTIONS:
Device: SETA LATECBA Stent Grafts — ABK model is a bifurcated polyester graft partially corrugated which is sutured at the proximal end (renal) to a balloon expandable 316 L stainless steel stent. The proximal half part of the stent is uncovered by polyester graft providing the anchoring to the healthy aorta wall when the device is implanted, as well as the perfusion of the renal arteries. The remaining half part is covered by polyester graft providing sealing of the aneurysm when it is expanded upon on the graft fabric and aneurysm neck. The distal end of each branch has the anchorage site for sealing after the connection with the iliac extensions RIK. The diameter of the anchorage site varies with the different ABK codes. The end of one branch is cone-shaped after the anchoring diameter with the purpose of promoting insertion of iliac extension RIK. The connection to iliac arteries is achieved by completing the aortic trunk ABK with 2 iliac extensions RIK.
  Other Names: ABK SETA LATECBA; RIK SETA LATECBA

SUMMARY:
This is a Prospective, Open-label, Multicenter, and Non-randomized Clinical Study. The main purpose of this study is to establish the efficacy and safety of a medical device system, SETA LATECBA Stent Graft, intended for the treatment of EVAR of pararenal AAA (patients with complex anatomy, not eligible for other surgical procedure).Other objective is to evaluate the technical performance of the device SETA LATECBA Stent Graft.

DETAILED DESCRIPTION:
This is a Prospective, Open-label, Multicenter, and Non-randomized Clinical Study to determine the Safety and Efficacy of the SETA LATECBA Stent Graft for endovascular repair therapy (EVAR) in Subjects with Abdominal Aortic Aneurysm (AAA)..The main purpose of this study is to establish the efficacy and safety of a medical device system, SETA LATECBA Stent Graft, intended for the treatment of Endovascular Aneurysm Repair (EVAR) of pararenal AAA (patients with complex anatomy, not eligible for other surgical procedure).

Secondary objective(s): The secondary objective is to evaluate the technical performance of the device SETA. LATECBA Stent Graft which includes: access to the implantation site, visualization, deployment of the stent- graft, sizing compatibility, withdrawal of the delivery system, and compatibility with ancillary equipment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults older than 18 years old, willing to cooperate with the study. No other demographic restriction.
* Initial diagnosis of AAA according to the standard of care criteria following the guidance Clinical Practice Guidelines for Endovascular Abdominal Aortic Aneurysm Repair
* Medical history: Complete history of previous, present and concomitant conditions, and current treatments for other conditions Signed informed consent. If the patient cannot consent, the subject's legally acceptable representative should consent

Diagnosis of Abdominal Aortic Aneurysm (AAA) according to the following criteria:

1. Diagnosis of an abdominal aortic aneurysm with a diameter ≥ 5.0 cm for males or ≥ 4.5 cm for females.
2. Aneurysm diameter with a growth rate ≥ 0.5 cm/ 6 months
3. The juxtarenal neck length between 1 mm and 10 mm
4. Neck diameter ≥16 to ≤ 26 mm
5. Suprarenal aorta diameter ≥ infrarenal aorta diameter
6. Proximal neck angulated ≤ 60 degrees relative to the long axis of the aneurysm
7. Immediate suprarenal aorta angulated ≤ 60 degrees relative to the immediate infrarenal neck.
8. Common iliac diameter 8 to 20 mm.
9. Common iliac length 25 mm
10. Common iliac angle 60 degrees
11. Not eligible for other standard EVAR surgical procedure

Exclusion Criteria:

* General Exclusion Criteria

  1. Life expectancy less than 2 years
  2. Pregnant or breastfeeding or planning on becoming pregnant within 60 months
  3. Included in another investigative drug or device study/studies or planning to do it within the following 24 months

Medical Exclusion Criteria

1. Previous treatment of AAA
2. Known allergy to polyester, stainless steel, nitinol and or gold, teflon, nylon,
3. Known anaphylactic reaction to contrast media.
4. Any type coagulopathy untreated.
5. Genetic connective tissue diseases, such as Marfan or Ehlers-Danlos syndromes
6. Planned interventional or surgical procedure within 30 days before or after AAA repair.
7. Renal dysfunction: creatinine level over 1.7 mg/dl
8. Systemic infection or fever over 38°C

   AAA Anatomy Exclusion Criteria
9. Significant occlusive disease, tortuosity, or calcification.

i) Significant thrombus in the fixation sites. j) Fungal aneurysm k) Leaking/ruptured or symptomatic aneurysm. l) Traumatic aneurysm. m) Concurrent aneurysm of the thoracic aorta. n) One or both renal arteries coming from the aneurysmal sac. o) Proximal neck diameter, measured outer wall to outer wall on a sectional image (CTA) > 26 mm in diameter or < 16 mm in diameter p) Proximal neck angle > 60 degrees relative to the long axis of the aneurysm q) Immediate suprarenal aorta angle > 60 degrees relative to the immediate infrarenal neck.

r) Immediate suprarenal aorta angle > 60 degrees relative to the immediate infrarenal neck s) Aortic diameter, measured inner wall to inner wall on a sectional image (CTA) < 15 mm at the bifurcation t) Iliac/femoral anatomy that is unsuitable for access. u) Iliac artery diameter, measured outer wall to outer Wall on a sectional image (CTA) > 20 mm or < 8 mm at distal fixation site.

v) Iliac artery distal fixation site < 10 mm in length. w) Indispensable inferior mesenteric artery (IMA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-12-11 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
EFFICACY: Number of participants with Endoleak Type I (measured by Angio CT Scan) | 30 days
  Type I endoleaks is diagnosed when there is a gap between the stent graft and the vessel wall. Usually is a result of the failure of the stent graft to achieve a circumferential seal of the aneurism. It produces systemic pressurization of the aneurysm sac and increases the risk of sac rupture.
SAFETY: mortality | 30-day
  percentage of died subjects

SECONDARY OUTCOMES:
SAFETY: Major Adverse Events | 30-day
  Composite endpoint including Q-wave myocardial infarction, Congestive heart failure, Cardiac ischemia requiring intervention Renal failure requiring dialysis, Bowel obstruction, ischemia or fistula, Stroke, Paralysis, Aneurysm leak and Device related death
Incidence of post-operative complications | 12 months
  Complications of aneurysm repair followed by secondary interventions
Clinical success | 30-day
  Composite endpoint including Successful deployment at intended site, No migration, Aneurysm exclusion, no type III and/or IV endoleak, No graft infection, No graft thrombosis, No aneurysm rupture, No conversion to open repair,
Clinical success | 6 months
  Composite endpoint including No migration, Aneurysm exclusion, no type I, III and/or IV endoleak, No graft thrombosis, No aneurysm rupture. No aneurysm diameter expansion >5 mm, No conversion to open repair
Clinical success | 12 months
  Composite endpoint including No migration, Aneurysm exclusion, no type I, III and/or IV endoleak, No graft thrombosis, No aneurysm rupture. No aneurysm diameter expansion >5 mm, No conversion to open repair
Technical Success of stent-graft implantation and delivery system usage | 12 months
  Composite endpoint including Assessment of system performance (Procedural times, Total blood loss, Deployment and device patency Ease of insertion, Visualization, Delivery system retrieval, Device integrity, Kinks, No type IV endoleak) Ancillary equipment needed, Adjunctive maneuvers (Balloon dilatation of aortic neck Balloon dilatation of iliac arteries, Additional stent or surgical procedure required, Eventual use of proximal cuff, Contrast media volume)

CONTACTS AND LOCATIONS:
Overall Officials: The-Bao Bui, MD, Principal Investigator — Centre Hospitalier Universitaire Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire Sherbrooke, Sherbrooke, Montreal, Canada

IPD SHARING:
Plan to Share IPD: No